CLINICAL TRIAL: NCT04360564
Title: Does a History of Recurrent Pregnancy Loss Predict a Prolonged Interval to the Second Live Birth or Increased Adverse Perinatal Outcomes for Women in British Columbia
Brief Title: RPL: Interval to Live Birth and Adverse Perinatal Outcomes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Children's & Women's Health Centre of British Columbia (Other)
Responsible Party: Principal Investigator, Dr. Mohamed Bedaiwy, Dr. Mohamed Bedaiwy, Professor in the Division of Reproductive Endocrinology & Infertility, Children's & Women's Health Centre of British Columbia
Other Study IDs: 1055
Record Dates: First submitted 2020-04-15; First posted 2020-04-24 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Abortion, Spontaneous; Abortion, Habitual; Birth Intervals; Pregnancy Loss; Pregnancy Complications
Keywords: recurrent pregnancy loss; time to live birth; live birth rate; perinatal outcomes
MeSH Terms: conditions — Abortion, Spontaneous; Abortion, Habitual; Pregnancy Complications

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Recurrent pregnancy loss: All women with >/=2 pregnancy loss before 20 weeks gestational age
  Interventions: Other: Recurrent pregnancy loss
- Primary recurrent pregnancy loss: Primary RPL is defined by those with >/=2 pregnancy loss before 20 weeks gestational age before the first birth
  Interventions: Other: Recurrent pregnancy loss
- Secondary recurrent pregnancy loss: Secondary RPL is defined by those with >/=2 pregnancy loss before 20 weeks gestational age occurring after the first birth
  Interventions: Other: Recurrent pregnancy loss
- No history of recurrent pregnancy loss: Those with 0 or 1 previous spontaneous pregnancy loss.

INTERVENTIONS:
Other: Recurrent pregnancy loss — As described before.
  Groups: Primary recurrent pregnancy loss; Recurrent pregnancy loss; Secondary recurrent pregnancy loss

SUMMARY:
This will be a retrospective observational cohort study utilizing the data from the British Columbia Perinatal Data Registry (BCPDR). The BCPDR is a provincially inclusive database that aggregates obstetrics and neonatal variables from all attended births in British Columbia.

The primary objective of this study is to evaluate and contrast the average time interval from the first to second birth for patients with recurrent pregnancy loss compared to healthy controls. Secondarily, the investigators will calculate the cumulative live birth rate in the cohort of women with recurrent pregnancy loss who were </= 35 at age of first birth and delivered between the years 2000-2010. Finally, the investigators will compare the incidence of adverse perinatal outcomes for those with recurrent pregnancy loss and those without.

The results of this study will be valuable for clinicians and patients as it will provide information for prognosis counselling. This will also help those desiring more than one child with long term family planning.

DETAILED DESCRIPTION:
Recurrent pregnancy loss (RPL) is defined as 2 or more pregnancy losses by the European Society of Human Reproduction and Embryology and affects 2-5% of the population. RPL can be further classified into primary and secondary pregnancy losses, with secondary RPL diagnosed when one has achieved a previous live birth. RPL is a frustrating and distressing condition as nearly 50% of patients have no medical explanation for the cause of pregnancy loss. For these patients, research regarding the prognosis and time to live birth is essential.

This will be a retrospective observational cohort study utilizing the data from the British Columbia Perinatal Data Registry (BCPDR). The BCPDR is a provincially inclusive database that aggregates obstetrics and neonatal variables from all attended births in British Columbia. Since April 2000, there are up to 700, 000 births included in this database. The study population will be divided into 4 groups: those without RPL (control group), all patients with RPL, primary RPL, and secondary RPL. Within the RPL group, primary RPL is defined by those with >/=2 pregnancy loss before 20 weeks gestational age before the first birth and the remaining patients will make up the secondary RPL group.

The following demographic variables will be requested: age at first delivery, age at second delivery, the average number of pregnancy loss before first birth, number of pregnancy loss before second birth, BMI at first delivery, BMI at second delivery, principle residence, use of in vitro fertilization to conceive, obstetrical status (number of pregnancies, term deliveries, preterm deliveries, miscarriages, and living children) at first and second birth, school years completed, smoking, at-risk alcohol use, preexisting hypertension, preexisting diabetes, psychiatric illnesses, the number of infant(s) born in first and second delivery, live birth/stillbirth. Primary outcome variables include the date (year, month, and day) of delivery for the first and second live births.

For our second objective, the investigators will analyze the cumulative live birth rate of a subgroup who is </= 35 at age of first birth and first delivery recorded between the year 2000-2010. The investigators will assume that this cohort will be more likely to try for a second pregnancy rather than an older group. Furthermore, there will be 10 to 20 years of follow-up data from the year 2010. A Kaplan-meier curve will be constructed showing the cumulative live birth rate for patients with RPL, primary RPL, secondary RPL, and control group, controlling for age, BMI, city of residence, use of IVF, number of miscarriages, consecutive RPL, and school years completed.

Lastly, the medical and obstetric characteristics of the pregnancies resulting in live birth after the diagnosis of RPL will be analyzed between the 4 groups (primary RPL, secondary RPL, all RPL, control). The associations between the previous diagnosis of RPL and adverse perinatal outcomes will be determined using logistic regression analyses.

ELIGIBILITY:
Inclusion Criteria:

* >/= 2 live births
* Livebirths occurring 2000-2020

Exclusion Criteria:

* Incomplete records
* Women with multiple gestations (at 1st or 2nd births)
* Stillbirths

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Those included in a provincially inclusive database that aggregates obstetrics and neonatal variables from all attended births in British Columbia from 2000-2018
Sampling Method: Non-Probability Sample
Enrollment: 140000 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Time between first birth and second birth | Time between first birth and second birth during 2000-2020
  Time interval in Weeks

SECONDARY OUTCOMES:
Live birth rate | 10 years after first live birth
  Proportion of patients achieving second live birth
Obstetrical outcomes | Live births during 2000-2020
  Gestational age at birth, antepartum hemorrhage, pregnancy-induced hypertension, intrauterine growth restriction, diabetes in pregnancy, mode of delivery, birth weight, maternal need for transfusion at delivery, sex of infant, APGAR at 5 and 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. Bedaiwy, FACOG, FRCSC, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital & Health Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho K, Fayek B, Liu YD, Albert A, Wiesenthal E, Dobrer S, AbdelHafez FF, Lisonkova S, Bedaiwy MA. A history of recurrent pregnancy loss is associated with increased perinatal complications, but not necessarily a longer birth interval: a population study spanning 18 years. Hum Reprod. 2024 May 2;39(5):1105-1116. doi: 10.1093/humrep/deae029. PMID 38390658